CLINICAL TRIAL: NCT00834080
Title: Open-Label Study of the Safety and Tolerability of VIVITROL Administered to Health Care Professionals Participating in an Extended Outpatient Treatment Program for Opioid Dependence
Brief Title: ALK21-021: A Safety Study of Medisorb® Naltrexone (VIVITROL®) Administered to Health Care Professionals
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALK21-021
Record Dates: First submitted 2009-02-02; First posted 2009-02-03 (Estimated); Results first posted 2013-07-29 (Estimated); Last update posted 2018-12-11 (Actual); Status verified 2018-11

CONDITIONS: Opiate Dependence
Keywords: opioid dependence; VIVITROL; opioid-related disorders
MeSH Terms: conditions — Opioid-Related Disorders | interventions — vivitrol; Naltrexone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Medisorb naltrexone 380 mg (VIVITROL) (Experimental)
  Interventions: Drug: Medisorb naltrexone 380 mg

INTERVENTIONS:
Drug: Medisorb naltrexone 380 mg — Intramuscular (IM) injection administered once every 4 weeks for up to 2 years
  Other Names: VIVITROL 380 mg; Naltrexone for extended-release injectable suspension

SUMMARY:
The purpose of this study is to determine the safety and tolerability of Medisorb® naltrexone (VIVITROL®) when administered over a period of 24 months to health care professionals who have a history of opioid dependence.

ELIGIBILITY:
Primary Inclusion Criteria:

* Health care professional (eg, physician, osteopath, nurse, pharmacist)
* 18 years of age or older
* Enrolled or enrolling in an extended outpatient treatment program for opioid dependence
* Women of childbearing potential must agree to use an approved method of contraception for the duration of the study

Primary Exclusion Criteria:

* Pregnancy and/or lactation
* Evidence of hepatic failure
* Active hepatitis
* Any psychiatric disorder that would compromise ability to complete study requirements
* Recent history of suicidal ideation or attempt
* Current dependence to any drugs other than prescription opioids or heroin, benzodiazepines, caffeine, marijuana, alcohol, or nicotine
* Positive urine drug test or self-reported use of opioids, cocaine, or amphetamines at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2009-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alkermes Medical Director, Study Director — Alkermes, Inc.
Locations (10):
- United States (10):
  - Alkermes Clinical Study Site, Colton, California
  - Alkermes Clinical Study Site, Oceanside, California
  - Alkermes Clinical Study Site, Lauderhill, Florida
  - Alkermes Clinical Study Site, Hoffman Estates, Illinois
  - Alkermes Clinical Study Site, St Louis, Missouri
  - Alkermes Clinical Study Site, Elmsford, New York
  - Alkermes Clinical Study Site, Canton, Ohio
  - Alkermes Clinical Study Site, Philadelphia, Pennsylvania
  - Alkermes Clinical Study Site, Austin, Texas
  - Alkermes Clinical Study Site, Dallas, Texas

REFERENCES:
- [Result] Earley PH, Zummo J, Memisoglu A, Silverman BL, Gastfriend DR. Open-label Study of Injectable Extended-release Naltrexone (XR-NTX) in Healthcare Professionals With Opioid Dependence. J Addict Med. 2017 May/Jun;11(3):224-230. doi: 10.1097/ADM.0000000000000302. PMID 28358754

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study had a 12 month recruitment period (May 2009 through April 2010). A total of 11 sites in the United States participated. Principal Investigators were addiction specialists who had contact with health care professionals in need of treatment for opioid dependence.
Pre-assignment Details: Potential subjects must have participated in a detoxification program for opioid dependence. Subjects participated in psychosocial treatment throughout their study participation.
Groups:
- VIVITROL: Study drug was administered by intramuscular (IM) injection once monthly for 24 months.
Period: Overall Study
Arm/Group | VIVITROL
Started | 38
Completed | 15
Not Completed | 23
Not completed — Adverse Event | 7
Not completed — Lost to Follow-up | 7
Not completed — Withdrawal by Subject | 5
Not completed — Other - Pregnancy | 1
Not completed — Other - False positive tests of the UDS | 1
Not completed — Physician Decision | 1
Not completed — Subject Relocated | 1

BASELINE CHARACTERISTICS:
Population: The Safety Population, defined as all subjects who received at least 1 dose (injection) of study drug, was used for presentation and analysis of both safety and efficacy data.
Arm/Group | VIVITROL, 380mg
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 38
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (10.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting at Least 1 Treatment-emergent Adverse Event (TEAE) While on Study.
Description: A TEAE is any adverse event (AE), whether or not considered drug-related, that develops or worsens in severity after study drug administration begins (ie, from the first administration through the end of the follow-up period).
Time Frame: 2 years (Baseline to end of study)
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | VIVITROL
Number analyzed (Participants) | 38
participants | 37

ADVERSE EVENTS:
Groups:
- Medisorb Naltrexone 380 mg (VIVITROL): Study drug was administered by intramuscular (IM) injection once monthly for 24 months.
Arm/Group | Medisorb Naltrexone 380 mg (VIVITROL)
Serious Adverse Events (participants affected / at risk) | 2/38
Other Adverse Events (participants affected / at risk) | 37/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medisorb Naltrexone 380 mg (VIVITROL) (N=38)
Head Injury (Injury, poisoning and procedural complications) | 1 (1)
Suicide Attempt (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medisorb Naltrexone 380 mg (VIVITROL) (N=38)
Injection site pain (General disorders) | 14 (25)
Fatigue (General disorders) | 4 (4)
Injection site induration (General disorders) | 3 (5)
Injection site mass (General disorders) | 3 (6)
Injection site nodule (General disorders) | 3 (3)
Irritability (General disorders) | 3 (3)
Chest pain (General disorders) | 2 (2)
Discomfort (General disorders) | 2 (3)
Oedema peripheral (General disorders) | 2 (3)
Pyrexia (General disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 16 (37)
Diarrhoea (Gastrointestinal disorders) | 5 (11)
Vomiting (Gastrointestinal disorders) | 5 (7)
Toothache (Gastrointestinal disorders) | 3 (6)
Abdominal discomfort (Gastrointestinal disorders) | 2 (6)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (3)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 11 (16)
Depression (Psychiatric disorders) | 5 (5)
Insomnia (Psychiatric disorders) | 3 (5)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 8 (9)
Bronchitis (Infections and infestations) | 5 (6)
Sinusitis (Infections and infestations) | 5 (6)
Tooth abscess (Infections and infestations) | 3 (5)
Urinary tract infection (Infections and infestations) | 3 (3)
Influenza (Infections and infestations) | 2 (3)
Headache (Nervous system disorders) | 10 (12)
Dizziness (Nervous system disorders) | 6 (6)
Amnesia (Nervous system disorders) | 2 (2)
Disturbance in attention (Nervous system disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 4 (8)
Increased appetite (Metabolism and nutrition disorders) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 3 (6)
Joint dislocation (Injury, poisoning and procedural complications) | 2 (2)
Muscle strain (Injury, poisoning and procedural complications) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Hypertension (Vascular disorders) | 2 (2)
Seasonal allergy (Immune system disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
After screening 49 subjects, Alkermes made a business decision to stop enrollment, resulting in 38 total subjects enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of such disclosure must be given to Alkermes for review at least sixty (60) days prior to submission for publication, presentation or delivery to any other party. Revisions to such disclosure will be negotiated in good faith by the Institution, Principal Investigator and Alkermes. Expedited reviews for abstracts or poster presentations may be arranged if mutually agreeable to Alkermes and the Institution.